CLINICAL TRIAL: NCT00532077
Title: An Exploratory, Open Label, Multicenter Parallel Group Study to Evaluate the Effects of Single and Repeat Dosing of SB-751689 (400 mg or 100 mg) or rhPTH(1-34) on the Fractional Renal Excretion of Calcium and Phosphate in Healthy Postmenopausal Females.
Brief Title: A Study to Evaluate the Effects of SB-751689 or rhPTH(1-34) on Excretion of Calcium and Phosphate in Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR9108122
Record Dates: First submitted 2007-09-17; First posted 2007-09-19 (Estimated); Last update posted 2010-10-19 (Estimated); Status verified 2010-10

CONDITIONS: Osteoporosis
Keywords: renal,; pharmacology,; Osteoporosis
MeSH Terms: conditions — Osteoporosis

INTERVENTIONS:
Drug: rhPTH(1-34)
Drug: SB-751689 100 mg
Drug: SB-751689 400 mg
  Other Names: rhPTH(1-34); SB-751689 100 mg

SUMMARY:
SB-751689 may alter calcium and phosphate handling at the kidney level. This study will examine what happens to calcium and phosphate, and other electrolytes, at the kidney after treatment with SB-751689 for 1 month. Another group of subjects will get another drug called Forteo for 1 month to compare the response of the kidney for calcium and phosphate.

ELIGIBILITY:
Inclusion Criteria:

* Healthy postmenopausal women 40 to 65 years of age, inclusive, meeting at least one of the following: Postmenopausal defined by the STRAW criteria of 12 months of spontaneous amenorrhea with serum FSH levels = 40 mIU/mL; History of bilateral oophorectomy (with or without hysterectomy) and at least 6 weeks post-surgical with serum FSH levels = 40 mIU/mL
* Body weight > 50 kg and BMI within the range 19 - 32 kg/m2
* Capable of giving written informed consent

Exclusion Criteria:

* Any clinically relevant biological or physical abnormality found or reported at screening which, in the opinion of the investigator, is clinically significant and would preclude safe participation in this study. These abnormalities may be identified on the screening history and physical or laboratory examination and 12-lead electrocardiogram (ECG).
* A subject may not participate in the study if any of the following laboratory results are above the upper limit of the normal range at screening: liver function tests (ALT, AST, GGT, alkaline phosphatase, total bilirubin), plasma amylase, glucose, alkaline phosphatase, or CPK.
* A subject may not participate in the study if any of the following laboratory results are outside the normal range at screening: serum levels of albumin-adjusted calcium, total calcium, PTH, and urinary calcium.
* A subject with vitamin D deficiency as defined by serum 25-hydroxy vitamin D < 20 ng/mL (equivalent to 50 nmol/L) at screening may not participate in the study. A QTc interval > 450 msec at screening.
* Positive urine drug screen.
* Positive for HIV, hepatitis B virus or hepatitis C virus assays.
* Urinary cotinine levels indicative of smoking.
* History of smoking or use of nicotine containing products within one year of screening.
* History of regular alcohol consumption
* History of drug abuse within 6 months of the study.
* Participation in a study with an investigational drug within 30 days or 5 half-lives (whichever is longer) preceding the first dose of study medication.
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, calcium containing antacids, aspirin or nonsteroidal anti-inflammatory drugs, vitamins, herbal and dietary supplements, excluding study related vitamin D and calcium supplements, within 14 days prior to the first dose of study medication.
* Donation of blood in excess of 500 mL within 56 days prior to dosing.
* Evidence of hepatic or biliary disease (including cholecystectomy and Gilbert's Syndrome).
* Significant renal disease as define by:
* Serum creatinine clearance <60ml/min (estimated from serum creatinine (SCr) and demographic data using the MDRD calculation):
* A validated web-based calculator is found at: http://nephron.com/cgi-bin/MDRDSIdefault.cgi
* GFR Calculator
* To calculate estimated GFR (mL/min/1.73m2) manually:
* = 186 x (SCr in mg/dL)-1.154 x (age)-0.203 x (0.742 if female) x (1.210 if African-American)
* = exp(5.228-1.154 x ln (SCr)-0.203x ln(age)-(0.299 if female) + (0.192 if African American))
* Urine protein/creatinine (mg/mg) ratio >2.5; or urine albumin concentration > 300 ug/mg.
* Known loss of kidney, either surgically or by injury or disease
* History of significant gastrointestinal
* History of a gastrointestinal surgical procedure that might affect the absorption of SB-751689
* History of sensitivity to any of the study medications or components thereof.
* History of clinically significant cardiovascular disease.
* History of pancreatitis or kidney stones. Medical conditions which might alter bone metabolism
* Subjects at increased risk of osteosarcoma such as those with Paget's disease of the bone or any prior external beam or implant radiation therapy involving the skeleton.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-08; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
renal fractional clearance of calcium and phosphate | over 1 month

SECONDARY OUTCOMES:
renal fraction clearance of electrolytes, cAMP, safety measures, and serum biomarkers | over 1 month
urinary excretion of sodium, magnesium, potassium, bicarbonate, and chloride
Albumin-adjusted serum calcium levels
Vitamin D and P1NP levels
Plasma levels of SB-751689 and rhPTH(1-34)
Plasma PTH
Adverse event reports, 12-lead ECGs, vital signs, nursing/physician observation and laboratory tests.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (5):
- United States (5):
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Daytona Beach, Florida
  - GSK Investigational Site, Port Orange, Florida
  - GSK Investigational Site, Honolulu, Hawaii
  - GSK Investigational Site, Austin, Texas